CLINICAL TRIAL: NCT04977557
Title: Efficacy of Thiamine in Patients With Clinically Suspected Dry Beriberi: An Open Labeled Hospital Bases Study in Bangladesh
Brief Title: Thiamine in Patients With Clinically Suspected Dry Beriberi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chittagong Medical College (Other)
Responsible Party: Principal Investigator, Nayema Masrura, Thesis Student, Department of Neurology, Chittagong Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 472
Record Dates: First submitted 2021-07-05; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Dry Beriberi
Keywords: Neuritic beriberi; Dry beriberi; thiamine efficacy
MeSH Terms: interventions — Thiamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): its a quasi experimental study where single group is used (self controlled clinical trial).
  clinical features were compared before iand after intervention
  Interventions: Dietary Supplement: Thiamine

INTERVENTIONS:
Dietary Supplement: Thiamine — Injection Thiamine 200 mg daily intravenously for 1 week followed by Tablet Thiamine 100mg bid for remaining 11 weeks

SUMMARY:
Abstract Background: Thiamine deficiency related disorders are increasingly being reported in countries where polished rice is the main dietary constituents and diet is not balanced in calorie, protein and micronutrients contents. Thiamine deficiency often associated with a sensory-motor neuropathy (dry beriberi) without Wernicke's encephalopathy and cardiac dysfunction.

Objectives: The objective of our study will be to evaluate the efficacy of thiamine in patients with clinically suspected dry beriberi.

Methods: This study will be a prospective, open labeled, self-controlled clinical trial (quasi-experimental study) carried out in the Neurology and Medicine Ward of Chittagong Medical College Hospital from July 2018 to June 2019. Fifty-five (55) patients of suspected dry beriberi will be recruited as per inclusion and exclusion criteria. All patients will be given 200mg IV Thiamine Hydrochloride per day for 1 week, then oral Tab. Thiamine 100mg twice daily for remaining 11week. They will be evaluated clinically before treatment and followed up at the end of 1 week, 6 week and 12 week after treatment. Assessment will be done by some clinical parameters like leg swelling, muscle cramp, muscle power, squat test, sensory impairments, deep tendon reflexes and by Overall Neuropathy Limitations Scale (ONLS) Score. Pre and post test treatment data will be recorded in a pre-designed case record form. To determine whether any o the difference between pretreatment and post treatment values were statistically significant or not, either Friedman's test or Cochran's Q test will be used. Analysis will be performed with SPSS windows version 23 and statistical significance will be defined as P<0.05 and confidence interval will be set at 95% level. Our study result is likely to sensitize the health professionals of this region about this neglected health issue by increasing awareness of the clinical spectrum of Thiamine Deficiency related Peripheral Neuropathy.

DETAILED DESCRIPTION:
This Self-controlled Clinical Trial will be conducted in Department of Neurology and Department of Medicine of Chittagong Medical College Hospital (CMCH) during July 2018 to June 2019. A total of 55 patients of possible beriberi will be included based on inclusion criteria. Patients with isolated cardiac/wet beriberi and with other known causes of peripheral neuropathy such as Diabetic, hereditary, Demyelinating (GBS, CIDP), metabolic (hepatic/renal impairment), history of intake of drugs (e.g. INH, Ethambutol, Phenytoin, Metronidazole, Dapsone etc.) and toxins exposure (As ,Organo-phosphate Compound, Pb ,Hg except alcohol) were excluded from study.

Operational Definitions:

Risk factors: Imbalanced diet (diet poor in thiamine/rich in carbohydrate or anti-thiamine factors), malnutrition, alcoholism, Gastro-Intestinal surgery, chronic diarrhoea, chronic vomiting, pregnancy or history of recent delivery, chronic, diuretics use, renal dialysis, total parenteral nutrition.

Possible/suspected neuritic (dry) beriberi: Risk factors + at least 2 of the following signs:

1. Muscle weakness of upper and or lower limb (less than grade 5 power in MRC scale)
2. Positive sensory symptoms (burning, tingling or pain)
3. Objective sensory deficit (pain, touch, position, vibration sense )
4. Absent or reduced deep tendon reflexes
5. Positive squat test (unable to rise after squatting without help)
6. Leg swelling Probable neuritic (dry) beriberi: Above symptoms recovered after thiamine treatment.

Data collection Procedure: After selection of subjects, detailed history, clinical examination and all other Information regarding sociodemographic and clinical factors of neuritic beriberi will be taken in a prescribed case record form. Relevant investigations (CBC, Peripheral Blood Flim (PBF), Serum creatinine, serum electrolytes, Liver function test, fasting & 2 hour after breakfast sugar. HbA1C, TSH, serum Vitamin B12, Chest X ray, ECG, Echocardiography, CSF study, Nerve Conduction Study will be performed to exclude differential diagnoses. Then therapeutic trial of Inj. Thiamine will be given IV for 1st week (200mg IV daily) then orally (tab. Thiamin 100mg bd) for 11 weeks. Patients will be followed up after 1, 6 and 12 week to see the response on the basis of some clinical parameters and Overall Neuropathy Limitations Scale (ONLS) score.

Statistical Analysis: Continuous data will be reported as the means ± SD or median and interquartile range. Qualitative or categorical data will be described as frequencies and proportions. The intention to treat analysis (ITT) analysis will be used to determine the statistical significance. Missing values will be replaced by the series means for this purpose. To determine whether any of the difference between pretreatment and post treatment values are statistically significant or not, either Friedman's test or Cochran's Q test will be used. Former test compares the quantitative variables and non-dichotomous qualitative variables and the later test compares the dichotomous qualitative/categorical variables. Statistical significance will be defined as P < 0.05 and confidence interval will be set at 95% level.

Variables under study:

Primary Outcome Variable: Treatment response will be measured by Overall Neuropathy Limitation Scale (ONLS) score before and after treatment.

Secondary Outcome Variables: Comparison and Assessment of clinical features at presentation and after treatment: leg swelling, muscle cramp, muscle power (MRC grading), deep tendon reflexes, sensory impairments (tingling /burning /pain/ touch/ position /vibration), squat test.

This study has received approval from Ethical Review Committee of Chittagong Medical College and written informed concent.will be taken from all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Any person admitted to CMCH as a Suspected thiamine deficiency related peripheral Neuropathy / Possible dry-beriberi:

   Risk factors + at least 2 of the following signs:

   Risk factors include Imbalanced diet (diet poor in thiamine/rich in carbohydrate or anti-thiamine factors), malnutrition, alcoholism, Gastrointestinal surgery, chronic diarrhoea, chronic vomiting, pregnancy or history of recent delivery, chronic. diuretics use, renal dialysis, total parenteral nutrition.
   1. Muscle weakness of upper and or lower limb (less than grade 5 power in MRC scale)
   2. Positive sensory symptoms (burning, tingling or pain)
   3. Objective sensory deficit (pain, touch, position, vibration sense )
   4. Absent or reduced deep tendon reflexes
   5. Positive squat test (unable to rise after squatting without help)
   6. Leg swelling
2. Age 18 years and above.

Exclusion Criteria:

1. Patients with isolated cardiac/wet beriberi.
2. Patient with known causes of peripheral neuropathy such as Diabetic, hereditary, Demyelinating (GBS, CIDP), metabolic (hepatic/renal impairment), drugs (e.g. Isoniazid, Ethambutol, Phenytoin, Metronidazole, Dapsone etc.) Toxin (As ,Organo-phosphate Compound (OPC), Pb ,Hg except alcohol) etc.
3. Patients refuse to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
change in Overall Neuropathy Limitation Scale (ONLS) score | before treatment with Thiamine (baseline ) and after 1 week, 6week, 12 week of treatment
  it is score measuring functional status of peripheral neuropathy patients. lowest score is 0 (No disability) and highest score 12 (most disability)

SECONDARY OUTCOMES:
change in leg swelling | before treatment with Thiamine (baseline ) and after 1 week, 6week, 12 week of treatment
  it may be mild (pitting disappears immediately after removing finger pressure), moderate (requiring less than 30 seconds to disappear after giving pressure), severe (requiring more than 30 seconds to disappear after giving pressure)
change in muscle power | before treatment with Thiamine (baseline ) and after 1 week, 6week, 12 week of treatment
  Medical Research Council (MRC) score is used, highest score 5 (Normal Power) and lowest score 0 (No muscle power)
change in muscle cramp | before treatment with Thiamine (baseline ) and after 1 week, 6week, 12 week of treatment
  Visual Analogue Scale (VAS) will be used for assessing severity of Muscle cramp. no cramp=0, mild cramp=1 to 3, moderate cramp= 4 to 6, severe cramp =7 to 10.
change in deep tendon reflexes | before treatment with Thiamine (baseline ) and after 1 week, 6week, 12 week of treatment
  deep tendon reflexes may be Normal , diminished or absent.
change in squat test | before treatment with Thiamine (baseline ) and after 1 week, 6week, 12 week of treatment
  squat test may be positive (inability or difficulty in raising from sitting position) or negative (no difficulty )
change in pain sensation | before treatment with Thiamine (baseline ) and after 1 week, 6week, 12 week of treatment
  Visual Analogue Scale (VAS) will be used for assessing severity of pain. no pain=0, mild pain= 1 to 3, moderate pain= 4 to 6, severe pain= 7 to 10.
change in position sensation | before treatment with Thiamine (baseline ) and after 1 week, 6week, 12 week of treatment
  it may be Normal , diminished or absent.
change in vibration sensation | before treatment with Thiamine (baseline ) and after 1 week, 6week, 12 week of treatment
  it may be Normal , diminished or absent.
change in touch sensation | before treatment with Thiamine (baseline ) and after 1 week, 6week, 12 week of treatment
  it may be Normal , diminished or absent.

CONTACTS AND LOCATIONS:
Overall Officials: Nayema Masrura, MD,MBBS, Principal Investigator — Thesis Student
Locations (1):
- Chittagong Medical College Hospital, Chittagong, Bangladesh

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT04977557/Prot_SAP_ICF_000.pdf